CLINICAL TRIAL: NCT05758974
Title: Postoperative Complications in Children Following Dental General Anesthesia and it's Correlation With The Type of Dental Treatment Done.
Brief Title: Postoperative Complication After G.A
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sawsan Ahmed Talaat, principal investigator in ministry of health,the health unit in Ibn betk fifth district in 6 October, Cairo University
Other Study IDs: complication of G.A
Record Dates: First submitted 2023-01-20; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Complication of Anesthesia
MeSH Terms: interventions — Dental Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: dental treatment — Extraction, pulp therapy or both

SUMMARY:
What are the possible postoperative complications that may occur for children following dental treatment under general anaesthesia and is there a correlation between those complications and type of dental treatment done?

DETAILED DESCRIPTION:
Nowadays, early childhood caries (ECC) remains a significant challenge of public health in Egyptian children. In most cases, children with ECC could accept dental treatment under non-pharmacological behavior management or sedation. However, some very young children or those suffering severe anxiety, mental or physical disabilities, could only be treated under dental general anesthesia (DGA).

Dental general anesthesia (DGA) is a safe and high-quality restorative and preventive treatment option for children with severe early childhood caries (S-ECC), who require extensive dental treatment and exhibit anxiety and emotional or cognitive immaturity or are medically compromised. However, several postoperative complications have been reported in children under DGA in many studies.

For a day-stay, general anesthesia procedure to be an acceptable option, care during and after surgery must be of the highest quality, and postoperative complications must be minimized.

ELIGIBILITY:
Inclusion Criteria:

1. Children with age range from 3 to 6 years old .
2. Children affected by dental caries in more than 4 primary teeth.
3. Uncooperative child indicated for treatment under G.A
4. Classified by American Society of Anaesthesiologists Physical Status as Class 1
5. Parents accepted to participate and willing to sign an informed consent.

Exclusion Criteria:

* 1) The children whose guardians or caregivers have a problem in communicating with the medical staff

Ages: 3 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: Children will be selected from general anaesthesia unit of Pediatric Dentistry Department, Faculty of Dentistry, Cairo University aged from 3-6 years according to the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-11-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Baseline
  pain would be assessed through the faces pain scale- revised this scale is self-report measure of pain intensity for children. These six faces expression show how much something can hurt, face 1 take score 0 no pain as minimum limit, face 2 take score 2, face 3 take score 4, face 4 take score 6, face 5 take score 8, face 6 take score 10 that the maximum limit "Very much pain."

SECONDARY OUTCOMES:
Fever | Baseline
  postoperative fever would be assessed through thermometer, the range of normal body temperature from (36,5 _37,5) °C. from (37,5- 38) ° Cit considers low grade fever. Above 38° C it considers high grade fever. Fever may be accompanied by irritable or very uncomfortable.
  poor eye contact with the surrounding, vomits repeatedly, severe diarrhea, seizures, pain.
  , severe headache, muscle weakness, difficulty breathing.
Weariness and drowsiness | Baseline
  That would be assessed through questionnaire.by asking the patient binary yes or no questions.

REFERENCES:
- [Background] Deng XY, Zhang YH, Zou J, Zhang Q. [Investigation of postoperative complications in children after dental therapy under general anesthesia]. Hua Xi Kou Qiang Yi Xue Za Zhi. 2020 Jun 1;38(3):284-289. doi: 10.7518/hxkq.2020.03.010. Chinese. PMID 32573136